CLINICAL TRIAL: NCT03238729
Title: Proof-of-Concept Study of a Smartphone Application Created to Improve Management of Ambulatory Patients With Heart Failure: the Heart Failure Heart Habits Application
Brief Title: Proof-of-Concept Study of Heart Habits Application for Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jana Care (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHF-MGH-001
Record Dates: First submitted 2017-07-28; First posted 2017-08-03 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHF App (Experimental): Patients will be provided with a mobile app on a smartphone for education and management of heart failure.
  Interventions: Behavioral: Heart Failure Education and Management App
- Standard of Care (Active Comparator): Patients will be provided standard literature on heart failure management.
  Interventions: Behavioral: Heart Failure Literature

INTERVENTIONS:
Behavioral: Heart Failure Education and Management App — Patients will be provided with an app on a smartphone that provides a daily checklist with items like reminders for logging weight and food, as well as educational components about heart failure and it's management.
  Arms: CHF App
Behavioral: Heart Failure Literature — Patients will be provided standard literature about heart failure and the management of heart failure.
  Arms: Standard of Care

SUMMARY:
This study assesses the ability of ambulatory patients with heart failure (HF) to use a smartphone application created for the management of patients with chronic HF. This study will aim:

* To understand the frequency with which ambulatory HF patients engage with this smartphone application.
* To determine whether patient's knowledge of HF and its management has improved with the use of this smartphone application.
* To assess improvement in quality of life measures related to the use of this smartphone application.
* To assess improvement in lifestyle measures related to the use of this smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HFrEF or HFpEF. HFrEF defined as clinical signs and symptoms of HF with a left ventricular (LV) EF ≤ 40% by any imaging modality AND at least 1 hospitalization or emergency department (ED) visit for HF or any outpatient escalation of diuretic therapy in the 12 months prior to study enrollment. HFpEF defined as clinical signs and symptoms of HF with an LVEF ≥ 50% by any imaging modality and at least 1 hospitalization or ED visit for HF or any outpatient escalation of diuretic therapy in the 12 months prior to study enrollment.
* Adult patients, men and women, > 18 years old.

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Number of patients that complete the curriculum | 6 weeks
  Total number of patients who complete the lessons on the app
Frequency of app use | 6 weeks
  Measuring how often and how long patients engaged with the app

SECONDARY OUTCOMES:
Score on Atlanta HF Knowledge Test | 6 weeks
  Assess patients knowledge of heart failure before and after study
Score on Kansas City Cardiomyopathy Questionnaire-12 | 6 weeks
  Assess changes in patients self-reported quality of life
%change in weekly activity as measured by steps | 6 weeks
  Assess changes in lifestyle measures (diet, activity, etc.)
Self reported frequency of weight measurement, exercise, fluid tracking, and sodium tracking | 6 weeks
  Compare baseline to end of study on a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hanna K Gaggin, MD, MPH, Principal Investigator — Massachusetts General Hospital; Nasrien E Ibrahim, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Konstam MA. Home monitoring should be the central element in an effective program of heart failure disease management. Circulation. 2012 Feb 14;125(6):820-7. doi: 10.1161/CIRCULATIONAHA.111.031161. No abstract available. PMID 22331919
- [Background] Gardetto NJ. Self-management in heart failure: where have we been and where should we go? J Multidiscip Healthc. 2011 Mar 31;4:39-51. doi: 10.2147/JMDH.S8174. PMID 21544247
- [Background] Powell LH, Calvin JE Jr, Richardson D, Janssen I, Mendes de Leon CF, Flynn KJ, Grady KL, Rucker-Whitaker CS, Eaton C, Avery E; HART Investigators. Self-management counseling in patients with heart failure: the heart failure adherence and retention randomized behavioral trial. JAMA. 2010 Sep 22;304(12):1331-8. doi: 10.1001/jama.2010.1362. PMID 20858878
- [Background] Shaw JD, O'Neal DJ 3rd, Siddharthan K, Neugaard BI. Pilot program to improve self-management of patients with heart failure by redesigning care coordination. Nurs Res Pract. 2014;2014:836921. doi: 10.1155/2014/836921. Epub 2014 Apr 23. PMID 24864206
- [Background] White MF, Kirschner J, Hamilton MA. Self-care guide for the heart failure patient. Circulation. 2014 Jan 21;129(3):e293-4. doi: 10.1161/CIRCULATIONAHA.113.003991. No abstract available. PMID 24446413
- [Background] Sochalski J, Jaarsma T, Krumholz HM, Laramee A, McMurray JJ, Naylor MD, Rich MW, Riegel B, Stewart S. What works in chronic care management: the case of heart failure. Health Aff (Millwood). 2009 Jan-Feb;28(1):179-89. doi: 10.1377/hlthaff.28.1.179. PMID 19124869
- [Background] Bonin CD, Santos RZ, Ghisi GL, Vieira AM, Amboni R, Benetti M. Construction and validation of a questionnaire about heart failure patients' knowledge of their disease. Arq Bras Cardiol. 2014 Apr;102(4):364-73. doi: 10.5935/abc.20140032. Epub 2014 Feb 17. PMID 24652054
- [Background] Masterson Creber RM, Maurer MS, Reading M, Hiraldo G, Hickey KT, Iribarren S. Review and Analysis of Existing Mobile Phone Apps to Support Heart Failure Symptom Monitoring and Self-Care Management Using the Mobile Application Rating Scale (MARS). JMIR Mhealth Uhealth. 2016 Jun 14;4(2):e74. doi: 10.2196/mhealth.5882. PMID 27302310
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL. 2013 ACCF/AHA guideline for the management of heart failure: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):1810-52. doi: 10.1161/CIR.0b013e31829e8807. Epub 2013 Jun 5. No abstract available. PMID 23741057
- [Background] WRITING COMMITTEE MEMBERS; ACC/AHA TASK FORCE MEMBERS. 2016 ACC/AHA/HFSA Focused Update on New Pharmacological Therapy for Heart Failure: An Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Card Fail. 2016 Sep;22(9):659-69. doi: 10.1016/j.cardfail.2016.07.001. Epub 2016 Jul 6. No abstract available. PMID 27394189
- [Background] Spertus JA, Jones PG. Development and Validation of a Short Version of the Kansas City Cardiomyopathy Questionnaire. Circ Cardiovasc Qual Outcomes. 2015 Sep;8(5):469-76. doi: 10.1161/CIRCOUTCOMES.115.001958. PMID 26307129
- [Background] Vieira AM, Costa IZ, Oh P, Lima de Melo Ghisi G. Questionnaires Designed to Assess Knowledge of Heart Failure Patients: A Systematic Review. J Cardiovasc Nurs. 2016 Sep-Oct;31(5):469-78. doi: 10.1097/JCN.0000000000000281. PMID 26208265
- [Background] Reilly CM, Higgins M, Smith A, Gary RA, Robinson J, Clark PC, McCarty F, Dunbar SB. Development, psychometric testing, and revision of the Atlanta Heart Failure Knowledge Test. J Cardiovasc Nurs. 2009 Nov-Dec;24(6):500-9. doi: 10.1097/JCN.0b013e3181aff0b0. PMID 19858959
- [Derived] Wei KS, Ibrahim NE, Kumar AA, Jena S, Chew V, Depa M, Mayanil N, Kvedar JC, Gaggin HK. Habits Heart App for Patient Engagement in Heart Failure Management: Pilot Feasibility Randomized Trial. JMIR Mhealth Uhealth. 2021 Jan 20;9(1):e19465. doi: 10.2196/19465. PMID 33470941